CLINICAL TRIAL: NCT06633042
Title: The Safety and Efficacy of Universal CAR-T Cells Targeting BCMA in the Treatment of Refractory AQP4 Antibody Positive Neuromyelitis Optica Spectrum Disease
Brief Title: The Safety and Efficacy of Universal CAR-T Cells Targeting BCMA in the Treatment of Refractory NMOSD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Wenzhou Medical University Affiliated Ophthalmology Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-BRL-302-01
Record Dates: First submitted 2024-09-25; First posted 2024-10-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Autoimmune Disease
Keywords: Universal BCMA CART; AQP4 Antibody Positive; RefractoryNeuromyelitis Optica Spectrum Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Total target count of CD3+CAR+ viable cells of 1E6/kg 、2E6/kg and 4E6/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART Group (Experimental): 1.0-4.0×10^6 CAR- Tcells/kg
  Interventions: Drug: Universal BCMA-CD19 CART

INTERVENTIONS:
Drug: Universal BCMA-CD19 CART — 1.0-4.0×10^6 CAR-T cells/kg
  Other Names: BRL-302

SUMMARY:
This is an open label, Multi-center，dose-escalation study in up to 18 participants with refractory NMOSD. This study aims to evaluate the safety and efficacy of universal CAR-T Cells targeting BCMA in the Treatment of refractory NMOSD.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label clinical study, and the sample size is set to 12-18 subjects. Based on the "3 + 3" dose escalation design principle, subjects will be divided into 3 groups from low dose to high dose in sequence (Group A; Group B; Group C).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years ; both genders eligible.
* Meets the criteria for Refractory NMOSD.
* Anticipated survival of ≥ 12 weeks as judged by the researcher.
* Agrees to use double barrier methods, condoms, oral or injectable contraceptives, or intrauterine devices during the study period and for one year after taking the study medication.
* Provides written informed consent.

Exclusion Criteria:

* History of solid organ transplantation.
* Malignant tumor within the last two years.
* Positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb), with peripheral blood Hepatitis B virus (HBV) DNA detected as positive; positive for Hepatitis C virus antibodies, with peripheral blood Hepatitis C virus RNA detected as positive; positive for Human Immunodeficiency Virus (HIV) antibodies; positive for Cytomegalovirus (CMV) DNA; positive for syphilis.
* Primary immunodeficiency (congenital or acquired).
* Severe cardiac disease.
* History of psychiatric disorders or history of psychotropic drug abuse, with no history of withdrawal.
* Allergic constitution or a history of severe allergies.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
DLT | Within28 Days After BRL-302 Infusion
  The number and severity of dose-limiting toxicity (DLT) events
AEs | Up to 12 Months After BRL-302 Infusion
  The total number, incidence, and severity of AEs

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) | 1,3,6,12 month after BRL-302 infusion
  Number of NMOSD relapses in subjects after cell infusion divided by observation time (years)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Wang, PhD, Study Chair — Wenzhou Medical University Affiliated Ophthalmology Hospital

IPD SHARING:
Plan to Share IPD: No